CLINICAL TRIAL: NCT04258917
Title: Impact of Crutch Type on Kinematics, Electromyography, Pain, and Comfort Following Knee Arthroplasty and Anterior Cruciate Ligament Reconstruction
Brief Title: Impact of Crutch Type on Gait and Functional Outcomes Post-knee Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemic prevented study from occuring
Sponsor: University of Calgary (Other)
Collaborators: University of Lethbridge (Other)
Responsible Party: Principal Investigator, Ranita Manocha, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0047
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Total Knee Arthroplasty; Anterior Cruciate Ligament Reconstruction
Keywords: crutches; gait; mobility; adult; knee replacement; ACL tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total Knee Arthroplasty (Experimental)
  Interventions: Device: Study withdrawn
- Anterior Cruciate Ligament Reconstruction (Experimental)
  Interventions: Device: Study withdrawn

INTERVENTIONS:
Device: Study withdrawn — Study withdrawn

SUMMARY:
Study withdrawn

DETAILED DESCRIPTION:
Study withdrawn

ELIGIBILITY:
Inclusion Criteria:

* Subjects 45-75 years old planning to get their first total knee replacement
* Subjects 18-45 years old planning to get their first anterior cruciate ligament reconstruction

Exclusion Criteria:

* Previous injury to shoulder, elbow, or wrist
* Current pain in shoulder, elbow, or wrist
* Inflammatory arthritis (i.e. rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis),
* History of cerebral palsy, stroke, significant cognitive impairment, or significant visual impairment
* Problems with the heart or lungs
* Currently using a crutch or crutches, walker, or other gait aid
* History of using a crutch or crutches for 4 or more weeks
* Inability to communicate in English
* Current smoker
* Currently pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Range of scapular downward rotation | Measured during gait assessment on post-operative day 4-12

SECONDARY OUTCOMES:
Bilateral upper extremity kinematics | Measured during gait assessment on post-operative day 4-12
  Hip flexion/extension, knee flexion/extension, and ankle dorsiflexion/plantar flexion; measured through optical motion tracking software
Bilateral upper extremity electromyographic (EMG) activity | Measured during gait assessment on post-operative day 4-12
Upper extremity pain | Measured at 3 time points: pre-operative, during gait assessment, and 4 weeks post-operative
  Measurements of pain at the shoulder, elbow, and wrist using an 11-point Numerical Rating Scale (0 = no pain, 10 = extreme pain)

OTHER OUTCOMES:
Weight-bearing lower extremity kinematics | Measured during gait assessment on post-operative day 4-12
  Hip flexion/extension, knee flexion/extension, and ankle dorsiflexion/plantar flexion; measured through optical motion tracking software
Torso kinematics | Measured during gait assessment on post-operative day 4-12
  Thoracic flexion/extension; measured through optical motion tracking software
Spatiotemporal parameters | Measured during gait assessment on post-operative day 4-12
  Gait velocity, crutch stride length, weight-bearing lower extremity stride length; measured through timing lights and computer software
Crutch comfort | Measured during gait assessment on post-operative day 4-12
  Measured through an 11-point Numerical Rating Scale for both crutch types (0 = extremely uncomfortable, 10 = extremely comfortable)
Number of falls | Measured at 4 weeks post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Ranita Manocha, MD, MSc, Principal Investigator — Department of Clinical Neurosciences, University of Calgary

IPD SHARING:
Plan to Share IPD: No